CLINICAL TRIAL: NCT01396889
Title: Impact of Echinacea as Prophilaxis for Upper Respiratory Tract Infections in Children 1-5 Years in Bandarabbas Children' Hospital
Brief Title: Impact of Echinacea as Prophilaxis for Upper Respiratory Tract Infections in Children 1-5 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hormozgan University of Medical Sciences (Other)
Responsible Party: Roya Firoozi, Hormozgan University of Medical Sciences (HUMS)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Echinacea in URIs
Record Dates: First submitted 2011-07-18; First posted 2011-07-19 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2010-05

CONDITIONS: Upper Respiratory Tract Infections
Keywords: Upper Respiratory Tract Infections; Echinacea; viral infections
MeSH Terms: conditions — Respiratory Tract Infections; Virus Diseases | interventions — Echinacea extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Echinacea (Experimental): 0.5ml daily for children 1-2 years old and 2ml daily for children2-5 years old for 3 months
  Interventions: Drug: Echinacea
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Echinacea — 0.5ml daily for children 1-2 years old and 2ml daily for children 2-5 years old
  Other Names: American Cone Flower
  Arms: Echinacea
Drug: Placebo — Placebo (0.5ml daily for children 1-2 years old and 2ml daily for children 2-5 years old) for 3 months
  Arms: Placebo

SUMMARY:
Acute upper respiratory tract infections are the most commmon infections in children and are associated with complications such as acute otitis media, sinusitis and pneumonia. Echinacea is widely used for treatment of upper respiratoty tract infections. The aim of this study is to evaluate its efficacy as prophilaxis in children 1-5 years old.

ELIGIBILITY:
Inclusion Criteria:

* Childrens 1-5 years old

Exclusion Criteria:

* Wheezing in previous 3 months requiring bronchodilatator
* History of hyperactive reactive airway
* using steroid or Echinacea
* chronic pulmonary of cardiac disease
* Acute respiratory disease within one week before study
* Allergic rhinitis
* Allergy to Echinacea
* avoiding to participate in the study

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2010-05; Primary Completion 2010-12 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
occurrence of upper respiratory tract infection diagnosed by physician according to history and physical examination and laboratory tests if was necessary | 6 months

SECONDARY OUTCOMES:
Drug side effects | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Roya Firoozi, Resident, Principal Investigator — Hormozgan University of Medical Sciences (HUMS)
Locations (1):
- Hormozgan University of Medical Sciences (HUMS), Bandar Abbas, Hormozgan, Iran